CLINICAL TRIAL: NCT01910025
Title: Phase 2 Study of ADI PEG 20 in Non-Hodgkin's Lymphoma Subjects Who Have Failed Prior Systemic Therapy
Brief Title: PH 2 ADI-PEG 20 Study in Non-Hodgkin's Lymphoma Subjects Who Have Failed Prior Systemic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2012-002
Record Dates: First submitted 2013-07-10; First posted 2013-07-29 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2016-04

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Argininosuccinate Synthetase; Arginine; Arginine deiminase; Failed prior systemic therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ADI PEG20; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental): arginine deiminase formulated with polyethlene glycol
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20
  Other Names: arginine deiminase formulated with polyethylene glycol

SUMMARY:
Certain cancers require the amino acid arginine. Arginine deiminase (ADI) is an enzyme from microbes that degrade arginine. ADI has been formulated with polyethylene glycol and has been used to treat patients that have cancers that have arginine. In this study, the primary efficacy variable will be assessment of tumor response rate.

ELIGIBILITY:
INCLUSION CRITERIA

1. Histologically proved NHL (B and T cells) according to WHO criteria and have relapsed or are refractory to at least 2 prior systemic chemotherapies (excluding chronic lymphocytic leukemia and Waldenstrom's macroglobulinemia).
2. Measurable disease as assessed by IHP criteria (Appendices A and B).
3. Age ≥ 20 years.
4. ECOG performance status of 0-2.
5. No prior systemic therapy, immunotherapy, investigational agent, or radiation therapy within the last 2 weeks prior to first dose of study treatment.
6. Fully recovered from any prior surgery and no major surgery within 4 weeks of initiating treatment. Surgery for placement of vascular access devices is acceptable.
7. Post-menarche female subjects and male subjects must be asked to use appropriate contraception for both the male and female for the duration of the study. Subjects must agree to use two forms of contraception or agree to refrain from intercourse for the duration of the study. Females must not be pregnant at the start of the study, and a serum human chorionic gonadotropin (HCG) pregnancy test must be negative before entry into the study.
8. Informed consent must be obtained prior to study initiation.
9. No concurrent investigational studies are allowed.
10. Absolute neutrophil count (ANC) >750/µL.
11. Platelets >50,000/µL.
12. Serum uric acid ≤ 8 mg/dL (with or without medication control).
13. Creatinine clearance must be ≥ 30 mL/min. This can be calculated using the Cockcroft-Gault equation: estimated creatinine clearance = [(140 - age) x weight (in kg)] / serum creatinine (in mg/dl) x 72; for females, multiple result by 0.85.

EXCLUSION CRITERIA

A subject will not be eligible for study participation if he/she meets any of the exclusion criteria:

1. Patients with infections requiring intravenous (IV) antibiotic/antiviral therapy are not eligible for entry onto the study; patients on prophylactic antibiotics or antivirals are acceptable.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.
5. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline (except alopecia) or ≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and investigator may be allowed upon agreement with both.
6. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current ASS negative cancer diagnosis.
7. Subjects who had been treated with ADI-PEG 20 previously.
8. History of seizure disorder not related to underlying cancer.
9. Known HIV positivity (testing not required).
10. Autologous or allogenic stem cell transplantation within 3 months before the first dose of study treatment.
11. Systemic steroids that have not been stabilized to the equivalent of ≧ 15 mg/day of prednisone 7 days prior to first dose of study treatment.
12. CNS lymphoma.
13. Allergy to pegylated compounds.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12-06 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Response Rate | 2 years estimated
  Determined by response criteria for cutaneous and non-cutaneous malignant lymphoma

SECONDARY OUTCOMES:
Safety and Tolerability | 2 years estimated
  Progression free survival - time from start of therapy until proven progression or death Overall survival Time on treatment Disease control rate Determine the pharmacodynamics of ADI-PEG 20 Determine the immunogenicity of ADI-PEG 20

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Chang Gung Medical Foundation-Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - CMUH, Taichung
  - National Cheng Kung University Hospital(NCKUH), Tainan
  - CGMH-LK, Taoyuan District